CLINICAL TRIAL: NCT06400940
Title: Prospective, Post-registration, Interventional, Randomized, in Parallel Groups, Multicenter Eurasian Clinical Study of DERIVO®/DERIVO® Mini Aneurysm Embolization Device, Europe-Asia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Andrey Evgenievich Petrov, MD, Principal Investigator, Head of Neurosurgical Department, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-ASIA
Record Dates: First submitted 2024-04-24; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Ticagrelor; Tablets; Prasugrel Hydrochloride; Aspirin

STUDY DESIGN:
Intervention Model Description: Prospective, post-registration, interventional, randomized, in parallel groups,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiplatelet (antithrombotic) monotherapy (Experimental): Antiplatelet (antithrombotic) monotherapy, including ticagrelor (tablets, 180 mg) or prasugrel (tablets, 10 mg).
  Interventions: Drug: ticagrelor (tablets, 180 mg) or prasugrel (tablets, 10 mg).
- Double antiplatelet (antithrombotic) therapy (Active Comparator): Double antiplatelet (antithrombotic) therapy (DAT), including a combination of clopidogrel (tablets, 75 mg) and acetylsalicylic acid (ASA, tablets, 100 mg) or a combination of ticagrelor (tablets, 180 mg) and ASA (tablets, 100 mg).
  Interventions: Drug: combination of clopidogrel (tablets, 75 mg) and acetylsalicylic acid (ASA, tablets, 100 mg) or a combination of ticagrelor (tablets, 180 mg) and ASA (tablets, 100 mg).

INTERVENTIONS:
Drug: ticagrelor (tablets, 180 mg) or prasugrel (tablets, 10 mg). — Antiplatelet (antithrombotic) monotherapy, including ticagrelor (tablets, 180 mg) or prasugrel (tablets, 10 mg).
  Arms: Antiplatelet (antithrombotic) monotherapy
Drug: combination of clopidogrel (tablets, 75 mg) and acetylsalicylic acid (ASA, tablets, 100 mg) or a combination of ticagrelor (tablets, 180 mg) and ASA (tablets, 100 mg). — Double antiplatelet (antithrombotic) therapy (DAT), including a combination of clopidogrel (tablets, 75 mg) and acetylsalicylic acid (ASA, tablets, 100 mg) or a combination of ticagrelor (tablets, 180 mg) and ASA (tablets, 100 mg).
  Arms: Double antiplatelet (antithrombotic) therapy

SUMMARY:
Prospective, post-registration, interventional, randomized, in parallel groups, multicenter Eurasian clinical study of DERIVO®/DERIVO® mini Aneurysm Embolization Device, Europe-Asia

DETAILED DESCRIPTION:
Prospective, post-registration, interventional, randomized, in parallel groups, multicenter Eurasian clinical study of DERIVO®/DERIVO® mini Aneurysm Embolization Device, Europe-Asia

ELIGIBILITY:
Inclusion Criteria:

* localization and structure of the aneurysm allows the use of a DERIVO®/DERIVO® mini flow-diverting stent for treatment;
* the aneurysm cannot be cured by other methods of endovascular therapy, or there is a higher risk of complications when using other methods of endovascular therapy or microsurgery;
* clipping or embolization with spirals (if performed earlier) led to a recurrence of the aneurysm.

Exclusion Criteria:

1. Age less than 18 years.
2. Pregnancy.
3. The presence of a previously implanted stent in a cerebral artery.
4. Dissection of cerebral or peripheral vessels.
5. The presence of contraindications to the use of the DERIVO®/DERIVO® mini medical device, specified in the instructions for use:

   * non-compliance of the aneurysm and/or the carrier vessel with the indications for the use of the device;
   * non-physiological structure of cerebral vessels;
   * vascular disorders that are a contraindication to endovascular interventions.
6. The presence of contraindications for antiplatelet (antithrombotic) and/or anticoagulant therapy in accordance with the instructions for the medical use of drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint: | For all participants from date of randomization and on visit 3 (3-6 months) and visit 4 study completion (12-18 months).
  The proportion of favorable clinical outcomes corresponding to 0-2 points on the modified Rankin Scale (mRS) for assessing clinical status in the medium-term (3-6 months) and long-term (12-18 months) postoperative period.

SECONDARY OUTCOMES:
Secondary endpoints: | For all randomized participants up to 2 weeks
  ● the proportion of technically successful stent implantations in the optimal position relative to the total number of treatment attempts using flow-diverting stents;
Secondary endpoints: | For all randomized participants up to 2 weeks
  ● the average amount of time required to install a flow-diverting stent;
Secondary endpoints: | baseline/discharge
  ● the change in the clinical status on the modified Rankin Scale (mRS) scale (0(no symptoms)-6 (death)) at the time of discharge compared with the value of the indicator at the screening.

OTHER OUTCOMES:
The technical success of stent implantation will be evaluated based on Digital subtraction angiography (DSA) on the fit of the flow-diverting stent to the wall of the carrier vessel according to the following criteria: | For all participants from date of randomization and on visit 3 (3-6 months) and visit 4 study completion (12-18 months).
  * proper fit of the device for deflecting the flow to the walls in the carrier vessel;
  * the gap between the flow deflection device and the vessel wall is < 25% of the vessel diameter;
  * the gap between the flow deflection device and the vessel wall is > 25% of the vessel diameter.
  * proper fit of the device for deflecting the flow to the walls in the carrier vessel;
  * the gap between the flow deflection device and the vessel wall is < 25% of the vessel diameter;
  * the gap between the flow deflection device and the vessel wall is > 25% of the vessel diameter.
  * proper fit of the device for deflecting the flow to the walls in the carrier vessel;
The technical success of stent implantation will be evaluated based on Digital subtraction angiography (DSA) on the fit of the flow-diverting stent to the wall of the carrier vessel according to the following criteria: | For all participants from date of randomization and on visit 3 (3-6 months) and visit 4 study completion (12-18 months).
  ● the gap between the flow deflection device and the vessel wall is < 25% of the vessel diameter;
The technical success of stent implantation will be evaluated based on Digital subtraction angiography (DSA) on the fit of the flow-diverting stent to the wall of the carrier vessel according to the following criteria: | For all participants from date of randomization and on visit 3 (3-6 months) and visit 4 study completion (12-18 months).
  ● the gap between the flow deflection device and the vessel wall is > 25% of the vessel diameter.
Clinical safety parameters: | through study completion, an average of 1,5 year
  ● the frequency of sensitivity to Double antiplatelet (antithrombotic) therapy or antiplatelet (antithrombotic) monotherapy according to the data of analyzer VerifyNow platelet testing and LTA platelet testing in patients of Mongoloid or Caucasoid races;
Clinical safety parameters: | through study completion, an average of 1,5 year
  ● the frequency of neurological disorders immediately after implantation of a flow- diverting stent;
Clinical safety parameters: | through study completion, an average of 1,5 year
  ● the frequency of bleeding and other AE caused by concomitant antithrombotic therapy;
Clinical safety parameters: | through study completion, an average of 1,5 year
  ● the frequency of acute cerebral circulation disorders in the medium-term (3-6 months) and long-term (12-18 months) postoperative period;
Clinical safety parameters: | through study completion, an average of 1,5 year
  ● frequency of deaths;
Clinical safety parameters: | through study completion, an average of 1,5 year
  the frequency of other Adverse Events and Serious Adverse Events
Angiographic safety parameters based on Digital subtraction angiography (DSA) | through study completion, an average of 1,5 year
  ● the frequency of complications associated with the intervention - stent opening, stent apposition to the vessel wall, thrombosis, thromboembolism, blockage of vascular branches affected by aneurysm.

CONTACTS AND LOCATIONS:
Locations (1):
- V.A. Almazov Fnmrc, Saint Petersburg, Russia